CLINICAL TRIAL: NCT02194907
Title: Emotion Study -- Improving Neural Dysregulation in Advanced Age: A Neurofeedback Approach
Brief Title: Emotion Study -- A Neurofeedback Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201300814 closed
Record Dates: First submitted 2014-07-10; First posted 2014-07-18 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Aging; Emotion
Keywords: Emotional Aging; Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior insula cortex activation (Active Comparator): Participants will receive training sessions using a special feedback technique to learn to actively increase blood flow in the front of the brain, while thinking of and viewing emotional faces, scenes, and text.
  Interventions: Behavioral: Brain activity training - anterior insula
- Primary auditory cortex activation (Active Comparator): Participants will have training sessions using a special feedback technique to learn to actively increase blood flow in the back of the brain while thinking of and viewing emotional faces, scenes, and text.
  Interventions: Behavioral: Brain activity training - medial prefrontal cortex

INTERVENTIONS:
Behavioral: Brain activity training - anterior insula — training sessions using a special feedback technique to learn to actively increase blood flow in the front of the brain
  Arms: Anterior insula cortex activation
Behavioral: Brain activity training - medial prefrontal cortex — training sessions using a special feedback technique to learn to actively increase blood flow in the back of the brain
  Arms: Primary auditory cortex activation

SUMMARY:
This study will determine whether brain activity can be modified and improves performance on a task by showing participants live 'video feed' of their brains on advanced imaging technology. The study is particularly interested in brain regions that have been shown to be relevant for emotions, specifically the anterior insula and the medial prefrontal cortex. Advanced technology will map the brain using magnetic pulses with a real-time functional Magnetic Resonance Imaging (rt-fMRI) machine.

DETAILED DESCRIPTION:
Overview: All participants of both age groups will be randomly divided (like tossing a coin) into two groups:

* One group will have training sessions using a special feedback technique to learn to actively increase blood flow in the front of the brain, while thinking of and viewing emotional faces, scenes, and text
* The other group will have training sessions using a special feedback technique to learn to actively increase blood flow in the back of the brain while thinking of and viewing emotional faces, scenes, and text

Further, each of these two groups will be divided into two sub-groups that are different with respect to the training procedure that is used:

* Use of a 3.0 Tesla, 32-channel Seimens whole-body human MR scanner (fMRI) during training, that has not been associated with any known side effects or safety risks

Number of Study Visits:

This study has the following parts: A pre-training visit, six training visits, and a post-training visit.

With a few exceptions as explained below, the procedures during pre-training, training, and post-training visits are identical.

* At the beginning of the first visit, the investigator will tell the participant about the study and what is involved and will ask them to sign a consent form. The participant may ask as many questions as they would like before deciding about study participation.
* For each of the visits, the investigator will review questions with the participant about their health to ensure their eligibility to undergo fMRI on the day of testing.
* Also for each visit, the investigator will ask the participant to respond to a short questionnaire related to their current mood.
* In the pre-training and the post-training visits only, the investigator will ask the participant to answer questions about their feelings, emotions, and thoughts.
* For each of the participant's visits, they will spend 50-60 minutes either in the MRI scanner, while viewing pictures and text on a screen. During this time, pictures of the participant's brain at work and at rest will be acquired. In the training visits only, the participant will learn to increase blood flow in certain brain regions with the help of information presented to them on the screen.
* For each of the participant's visits, they will be asked to respond to a short questionnaire related to their current mood.
* In the pre-training/post-training visits only, the investigator will ask the participant to answer questions about their feelings, emotions, and thoughts as well as their personality. The participant will also perform brief tests related to the thinking process.
* At the end of each visit, the participant will complete a questionnaire about how they approached the study tasks and whether they experienced any discomfort in the MRI scanner or while wearing the fNIRS system.
* Upon study completion, the investigator will tell the participant about the general goals of the study and answer any questions that they may have.

The procedure can be stopped at any time.

The study will conclude with debriefing and reimbursement.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30 years or 63-90 years
* Right-handed
* Native English speaker

Exclusion Criteria:

* Pregnant or possibly pregnant
* Claustrophobia
* Large pieces of metal in the body, particularly in the face and neck.
* Piercings or metal implants that cannot be removed from the body
* Surgery on the brain or any prior serious brain damage or disease
* Dementia or severe cognitive disorders

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-10; Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Increased activation of anterior insula from pre-training to post-training | Pre-training session (baseline visit); post-training session (approximately one week later)
  Both young and older participants can be trained in up-regulation of anterior insula activity, by means of contingent neurofeedback (rt-fMRI), reflecting continued plasticity of brain regions associated with affective processing.

SECONDARY OUTCOMES:
Gained volitional control over activity in anterior insula improves emotion perception from pre-training to post-training | Pre-training (baseline visit); post-training visit (approximately one week later)
  Participants in the experimental group compared to the control group will benefit more from neurofeedback, in that they will show relatively greater improvement in emotion perception after the rt-fMRI training, reflecting a potential for improvement of neural dysregulation related to affective processing.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Ebner, PhD, Principal Investigator — University of Florida, Department of Psychology
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- See also: Real-Time fMRI in Neuroscience Research and Its Use in Studying the Aging Brain — http://www.frontiersin.org/articles/10.3389/fnagi.2016.00239/full